CLINICAL TRIAL: NCT00793650
Title: Combination High Dose Melphalan and Autologous PBSC Transplant With Bortezomib for Multiple Myeloma: A Dose and Schedule Finding Study
Brief Title: Combination High Dose Melphalan and Autologous Peripheral Blood Stem Cell (PBSC) Transplant With Bortezomib for Multiple Myeloma: A Dose and Schedule Finding Study
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Sagar Lonial, MD, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 080-2005
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2012-06-18 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Cancer; Multiple Myeloma
Keywords: Cancer; Multiple Myeloma; Peripheral Blood Stem Cell Transplant
MeSH Terms: conditions — Neoplasms; Multiple Myeloma | interventions — Bortezomib; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bortezomib before Melphalan (Active Comparator): Enrolled patients were randomized to receive a single escalating dose of bortezomib (1.0, 1.3, or 1.6 mg/m2) 24 hours before melphalan.
  Interventions: Drug: Bortezomib; Drug: Melphalan; Procedure: Autologous PBSC Transplant
- Bortezomib after Melphalan (Active Comparator): Enrolled patients were randomized to receive a single escalating dose of bortezomib (1.0, 1.3, or 1.6 mg/m2) 24 hours after melphalan.
  Interventions: Drug: Bortezomib; Drug: Melphalan; Procedure: Autologous PBSC Transplant

INTERVENTIONS:
Drug: Bortezomib — Escalating doses of bortezomib 1.0, 1.3, or 1.6 mg/m2 in Arm A and Arm B.
  Other Names: Bortezomib or Velcade
Drug: Melphalan — All patients received melphalan (100 mg/m^2/day × 2; days
  -3 and -2), for a total dose of 200 mg/m^2.
  Other Names: Bortezomib or Velcade
Procedure: Autologous PBSC Transplant — Day 0 consists of the stem cell infusion.

SUMMARY:
The goal of this study is to evaluate the safety of melphalan and autologous PBSCT (peripheral blood stem cell transplantation - stem cells that come from your own body) in combination with bortezomib, a new FDA approved drug used to treat myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma who are eligible for an autologous peripheral blood progenitor transplant
* Male and female subjects between the age of 18 and 70 years.
* Patient has given informed consent prior to any study related procedures with the knowledge that consent can be withdrawn at anytime without prejudice to future medical care
* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subjects agrees to use an acceptable method for contraception for the duration of the study.
* Biopsy proven diagnosis of multiple myeloma from bone marrow aspirate and biopsy prior to study initiation
* Patient has achieved less than 90% disease reduction from previous treatment prior to transplant (as measured by serum or urine protein electrophoresis) and has more than 5% plasma cells in the bone marrow, or patient has progressed and has more than 5% plasma cells in the bone marrow.
* Karnofsky Performance Status score of ≥ 60%
* Patient has met the following laboratory requirements prior to Day -4
* Platelet count ≥ 50, 000/mm3
* Absolute Neutrophil Count ≥ 500/mm3
* Hemoglobin ≥ 10 g/dL (transfusion allowed to meet this criterion)
* Calculated creatinine clearance ≥ 30mL/min
* Toxic effects of previous therapy or surgery resolved to Grade 2 or better

Exclusion Criteria:

* Unsupportable anemia with < 10b/dL
* Patient has a calculated or measured creatinine clearance of < 30mL/min within 14 days before enrollment
* Patient has ≥ Grade 2 peripheral neuropathy within 14 days before enrollment
* Patient has hypersensitivity to bortezomib, boron or mannitol
* Patient has had an allergic reaction to melphalan or chlorambucil
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Cardiac or pulmonary dysfunction such that patients do not meet institutional pre-transplant evaluation criteria
* Known central nervous system involvement or suspicion of involvement with Myeloma
* Other active malignancies (with the exception of basal and squamous cell skin cancer) within 5 years of study entry. Patients with treated prostate or cervical cancer in situ who are 2 or more years from therapy and remain free of disease may be entered into the study at the investigator's discretion.
* Known to be HIV positive, HIV-1 positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-05; Primary Completion 2009-10 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Lonial, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib Before HD Melphalan: All patients received melphalan (100 mg/m^2/day × 2; days
  -3 and -2), for a total dose of 200 mg/m^2. Patients were randomized to receive bortezomib 24 hours before administration of high-dose melphalan in escalating dose cohorts of 1.0, 1.3, and 1.6 mg/m^2
- Bortezomib After HD melphalanAll: patients received melphalan (100 mg/m^2/day × 2; days
  -3 and -2), for a total dose of 200 mg/m^2. Patients were randomized to receive bortezomib 24 hours after administration of high-dose melphalan in escalating dose cohorts of 1.0, 1.3, and 1.6 mg/m^2
Period: Overall Study
Arm/Group | Bortezomib Before HD Melphalan | Bortezomib After HD melphalanAll
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bortezomib Before HD Melphalan | Bortezomib After HD melphalanAll | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 5 | 6 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 58.32 (7.92) | 58.75 (8.05) | 58.54 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Safety and Engraftment
Description: Peripheral blood progenitor cells were collected with either chemo-mobilization (27 of 39, 69%) or growth factor mobilization (12 of 39, 31%). Patients received an average of 9.0 × 10^6/kg CD34+ cells (range, 2.3-65) as their transplant graft.
Time Frame: Day 30 after transplant
Population: As per the protocol
Measure: Median (Full Range); unit: days
Arm/Group | Bortezomib Before HD Melphalan | Bortezomib After HD melphalanAll
Number analyzed (Participants) | 19 | 20
days
  Median time for platelet recovery | 16 [8 to 23] | 16 [10 to 58]
  Median time for neutrophil recovery | 12 [10 to 18] | 12 [9 to 35]

2. Secondary Outcome: Response Rate Using EBMT(European Group for Blood and Bone Marrow Transplan) Criteria at Day +100 After Transplant.
Description: CR :Negative immunofixation on the serum and urine and Disappearance of any soft tissue plasmacytomas and <=5% plasma cells in bone marrow.
  VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100mg per 24 hour.
  Partial Response:>=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200mg per 24 hour.
Time Frame: 100 days after transplant
Population: As per the protocol.
Measure: Number; unit: participants
Groups:
- Bortezomib Before Melphalan: All patients received melphalan (100 mg/m^2/day × 2; days
  -3 and -2), for a total dose of 200 mg/m^2. Patients were randomized to receive bortezomib 24 hours before administration of high-dose melphalan in escalating dose cohorts of 1.0, 1.3, and 1.6 mg/m^2
- Bortezomib After Melphalan: patients received melphalan (100 mg/m^2/day × 2; days
  -3 and -2), for a total dose of 200 mg/m^2. Patients were randomized to receive bortezomib 24 hours after administration of high-dose melphalan in escalating dose cohorts of 1.0, 1.3, and 1.6 mg/m^2
Arm/Group | Bortezomib Before Melphalan | Bortezomib After Melphalan
Number analyzed (Participants) | 19 | 20
participants
  Complete response (CR) | 2 | 6
  VGPR-Very good partial remission | 9 | 11
  Partial Response | 6 | 7

ADVERSE EVENTS:
Arm/Group | Bortezomib Before HD Melphalan | Bortezomib After HD melphalanAll
Serious Adverse Events (participants affected / at risk) | 4/19 | 2/20
Other Adverse Events (participants affected / at risk) | 19/19 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib Before HD Melphalan (N=19) | Bortezomib After HD melphalanAll (N=20)
Expired (General disorders) | 3 | 1
Acute pulmonary embolus (General disorders) | 0 | 1
Hemorrhage/Bleeding-Hemorrhage (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib Before HD Melphalan (N=19) | Bortezomib After HD melphalanAll (N=20)
Muscositis (Gastrointestinal disorders) | 18 | 16
Diarrhea (Gastrointestinal disorders) | 16 | 18
Nausea (Gastrointestinal disorders) | 19 | 18
Vomiting (Gastrointestinal disorders) | 11 | 11
Febrile Neutropenia (Blood and lymphatic system disorders) | 11 | 13
Sepsis (Infections and infestations) | 3 | 2
Liver Toxicities (Hepatobiliary disorders) | 5 | 4
Clostridium diificile (Gastrointestinal disorders) | 3 | 1
Renal toxicities (Renal and urinary disorders) | 4 | 7
Rash (Skin and subcutaneous tissue disorders) | 2 | 5
Cognitive disturbances (Nervous system disorders) | 2 | 1
Seizures (Nervous system disorders) | 1 | 0
DVT/PE (Vascular disorders) | 1 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0
Hypernatremia (General disorders) | 2 | 1
Headaches (General disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pulmonary toxicities (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Incontinenece (Renal and urinary disorders) | 1 | 0
Gastrointestinal bleed (Gastrointestinal disorders) | 1 | 0
Neutopenic colitis (Gastrointestinal disorders) | 0 | 1
Blisters on Feet (Skin and subcutaneous tissue disorders) | 1 | 0
Urinary retension (Renal and urinary disorders) | 0 | 1
Hypotension (Cardiac disorders) | 4 | 2
A.fib (Cardiac disorders) | 1 | 0
sinus bradycardia (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes